CLINICAL TRIAL: NCT02856074
Title: Prognosis After Revascularization Therapy in the Dijon Ischemic Stroke Evaluation Study
Brief Title: Functional Prognosis in Patients With Ischemic Stroke According to the Therapeutic Strategy Used
Acronym: PARADISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Béjot 2015-2
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

ARMS (1):
- Ischemic stroke patients (Experimental)
  Interventions: Biological: prise de sang; Other: quality of life questionnaire

INTERVENTIONS:
Biological: prise de sang
Other: quality of life questionnaire

SUMMARY:
The current management of ischemic stroke is based on different strategies that may be combined: intravenous thrombolysis in a stroke ICU, intravenous thrombolysis in a telemedicine procedure, endovascular thrombectomy. Given this now rich therapeutic arsenal, it seems necessary to evaluate practices in local care in the field and the impact of these on the prognosis of ischemic stroke victims. The aim of this observational study is to compare these different care practices without interfering with the choice of strategy.

A blood sample will also be taken at different times to study the value of growth differentiation factors (GDF) 8, 11 and 15, and Brain-derived Neurotrophic Factor as prognostic biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic ischemic stroke defined according to WHO criteria and treated by intravenous thrombolysis at the stroke ICU at Dijon CHU, intravenous thrombolysis by telemedicine with subsequent transfer to the Dijon stroke ICU, and/or endovascular thrombectomy at Dijon CHU)
* Patients aged over 18 years.
* Patients who have provided written informed consent to take part in the study.

Exclusion Criteria:

* Patients who refuse to take part in the study.
* Subjects in custody.
* Patients (or a person of trust) who cannot be contacted by telephone during the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of handicap | 6 months

SECONDARY OUTCOMES:
Serum levels of biomarkers of stress | Changes compared with baseline levels at Day 1, Day 3, Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France